CLINICAL TRIAL: NCT06448403
Title: Multimodal Assessment of Cognitive Impairment in Alzheimer Patients
Brief Title: Multimodal Assesment of Alzheimer Patients
Acronym: MultiAD
Status: Recruiting | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 626476
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease, Late Onset; Cognitive Impairment; Dementia
Keywords: Alzheimer Disease (AD); Mild cognitive impairment (MCI); Brain Diseases; Nervous System Disorders; Neurodegenerative Diseases; Dementia; Cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia; Brain Diseases; Nervous System Diseases; Neurodegenerative Diseases | interventions — Polysomnography; Blood Specimen Collection; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MCI: Recruitment according to relevant clinical assessment and ICD-criterias.
  Interventions: Device: MRI Scanning; Device: 64-channel EEG; Device: Polysomnography; Biological: Blood samples; Biological: Fecal samples; Behavioral: Cognitive tests
- Mild AD: Recruitment according to relevant clinical assessment and ICD-criterias.
  Interventions: Device: MRI Scanning; Device: 64-channel EEG; Device: Polysomnography; Biological: Blood samples; Biological: Fecal samples; Behavioral: Cognitive tests
- Control: Equivalent number of research participants as in the MCI and mild AD group.
  Interventions: Device: MRI Scanning; Device: 64-channel EEG; Device: Polysomnography; Biological: Blood samples; Biological: Fecal samples; Behavioral: Cognitive tests

INTERVENTIONS:
Device: MRI Scanning — MRI scanning with volumetric, resting and activity-based sequences.
Device: 64-channel EEG — EEG to quantifiy electric activity.
Device: Polysomnography — A randomized group will undergo polysomnography.
Biological: Blood samples — Analysis of specific blood biomarkers.
Biological: Fecal samples — Analysis of bacterial composition.
Behavioral: Cognitive tests — Interview-based cognitive tests for assesment of cognitive levels.

SUMMARY:
The goal of this study is to learn more about the changes in the brains of patients with cognitive impairment (MCI) and Alzheimer's Disease (AD).

The main questions the study aims to answer are:

1. What findings can be used to earlier detect patients that will develop Alzheimers?
2. Which differences are seen between healthy and cognitively impaired patients?
3. Which differences are seen between patients with Alzheimers disease?

Participants will undergo:

* Cognitive tests
* Magnetic resonance imaging (MRI)
* Electroencephalography (EEG)
* Blood sample collection
* Fecal sample collection
* A randomized group will undergo polysomnography analysis.

DETAILED DESCRIPTION:
The projects aims to map brain changes in patients with mild cognitive impairment (MCI) and Alzheimer's Disease (AD) by combining different assesment modalities.

In the MRI, researchers will get the opportunity to analyse both structural and functional brain changes. In the EEG, changes in elctrical activites will be measured. The blood samples allow researchers to analyse specific dementia and inflammation proteins, while fecal speciments can be used to assess bacterial composition. Additionally, the cognitive testing allow to assess the specific part of cognitive function which is affected.

ELIGIBILITY:
Inclusion Criteria:

* MCI and AD according to relevant ICD-criterias.
* Control cohort is age and gender matched with other cohorts.

Exclusion Criteria:

* Uneligibility for any of the planned neuroimagery devices (MRI, EEG)
* AD diagnosis before the age of 65 (Early-onset AD).
* Brain tumor
* Traumtic head injury
* Earlier neurosurgery
* Other neyrodegenerative diseases (i.e Parkinson and ALS)
* Diseases related to inflammation and auto-immunity (i.e MS)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study population is from Tronderlag in Norway, mainly in and around Trondheim city.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2030-12-29 (Estimated); Study Completion 2030-12-29 (Estimated)

PRIMARY OUTCOMES:
MCI-AD converters | 5 years
  Identify biomarker profiles unique for patients with MCI that develop AD for earlier prediction.
AD-subclassification | 5 years
  Identify biomarker profiles that can assist in a more thorough AD-classification

CONTACTS AND LOCATIONS:
Overall Officials: Axel Sandvig, Prof., MD, PhD, Principal Investigator — Norwegian University of Science and Technology (NTNU) & St. Olavs Hospital, Trondheim University Hospital
Locations (1):
- Norwegian University of Sciene and Technology / Norges teknisk-naturvitenskapelige universitet (NTNU), Trondheim, Trønderlag, Norway